CLINICAL TRIAL: NCT00387192
Title: An Open Multi-centre Study in Patients With Von Willebrand Disease to Investigate the Pharmacokinetics, Efficacy and Safety of OPTIVATE®, a High Purity, Dual Inactivated Factor VIII and Von Willebrand Factor Concentrate
Brief Title: A Study With OPTIVATE® in People With Von Willebrand Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to slow recruitment and a significant delay in reaching the recruitment target.
Sponsor: Bio Products Laboratory (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8VWF01
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-03

CONDITIONS: Von Willebrand Disease
Keywords: Von Willebrand Disease; Factor VIII; Von Willebrand Factor; Pharmacokinetics
MeSH Terms: conditions — von Willebrand Diseases; Hemophilia A | interventions — optivate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Optivate — Plasma-derived Factor VIII

SUMMARY:
The main objective of the study is to assess the pharmacokinetics of OPTIVATE® after a single dose of 80 IU/kg VWF:RCo. The secondary objectives of the study are to assess efficacy and safety of OPTIVATE® in long-term use over at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent.
2. Be aged 12 years or older.
3. Have severe VWD (VWF:RCo <20%) of known type. Severity will be confirmed by a current VWF:RCo result of <20%.
4. Be known or expected to require a concentrate for management of VWD.
5. Must have had at least one bleed in the last 12 months which required treatment with a FVIII and VWF concentrate.
6. Have a known lack of, or poor response to, DDAVP.
7. Have a prothrombin time (PT) of not more than 3 seconds above the upper limit of the reference range.
8. At the Baseline Visit (Visit 1), patients must have had at least 5 days since their last infusion of replacement factor concentrate or DDAVP.
9. Female patients of child-bearing potential must have a negative result on a human chorionic gonadotropin-based pregnancy test. If a female patient is or becomes sexually active, she must practice contraception by using a method of proven reliability for the duration of the study. Female patients must not be lactating.

Exclusion Criteria:

1. Have a history of inhibitor development to VWF or FVIII or a positive result at screening.
2. Actively bleeding (Note: the patient can enter the study once the bleed is controlled).
3. Presence of major systemic illnesses: renal disease, liver disease, or neurological or psychiatric disease which would compromise the outcome of the study in the opinion of the investigator.
4. Known or suspected hypersensitivity to investigational medicinal product (IMP) or its excipients.
5. Have a recent history of alcohol or drug abuse.
6. Administration of a new chemical entity within the 4 months preceding enrolment.
7. Participation in any other clinical study in which investigational or marketed drugs were employed in the 30 days preceding enrolment into this study, with the exception of the BPL clinical study Protocol 8VWF03.
8. In the opinion of the investigator, the patient is unlikely to comply with the study protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2006-11; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters for VWF RCo at the Baseline Visit by VWD type and overall. | Baseline vist

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hay, MD, Principal Investigator — Manchester Haemophilia Comprehensive Care Centre
Locations (4):
- Israel (3):
  - Rambam Health Care Campus, 8 Haaliya St., Bat-Galim, Haifa
  - Haddasah Ein-Karem Medical Center, P.O.Box 12000, Jerusalem
  - Beilinson Hospital, Rabin Medical Center, 39 Jabontinsky Street, Petah Tikva
- University Department of Haematology, Manchester, United Kingdom

REFERENCES:
- See also: Sponsor's homepage — http://www.bpl.co.uk